CLINICAL TRIAL: NCT02866552
Title: SCLERoderma et Adipose-DErived Stroma Cells
Acronym: SCLERADECIII
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2016-40
Record Dates: First submitted 2016-08-05; First posted 2016-08-15 (Estimated); Last update posted 2016-08-15 (Estimated); Status verified 2016-08

CONDITIONS: Systemic Sclerosis
MeSH Terms: conditions — Scleroderma, Systemic | interventions — Ringer's Lactate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PLACEBO (Placebo Comparator): Patients will receive an injection of placebo
  Interventions: Drug: Ringer lactate
- DRUG : Stromal Vascular Fraction (Experimental): Patients will receive an injection of Stromal Vascular Fraction injection
  Interventions: Drug: Stromal Vascular fraction

INTERVENTIONS:
Drug: Stromal Vascular fraction
  Arms: DRUG : Stromal Vascular Fraction
Drug: Ringer lactate
  Other Names: placebo
  Arms: PLACEBO

SUMMARY:
Systemic sclerosis (SSc) is an auto-immune orphan disease mainly characterized by an alteration of the microvascular network, and by cutaneous and visceral fibrosis. Hands are frequently affected, as a consequence of ischemic phenomena and cutaneous fibrosis. As a result, patients suffer from everyday disability, with consequences on their occupational activities and social contact, sometimes severely altering their quality of life. To date, no anti-fibrosis treatment has proven effective; existing vasodilation treatments are unfortunately not very effective, and are associated with adverse effects or restrictions. It is consequently of utmost importance that an effective treatment for sclerodermic hands be developed. The injection of adipose autologous tissue is a common practice in plastic surgery, and has been known for over a century. Adipose tissue, originally used to increase volume, is also characterized by trophic properties associated to stromal vascular fraction (SVF), which contain multipotent stem cells, capable of tissue repair. Interestingly, some SVF cells can be angiogenic and anti-inflammatory, which could improve damage seen with SSc. The injection of SVF into the fingers would also make it possible to control the production of the extracellular matrix and to improve the balance between fibrosis and fibrolysis, resulting in an improvement of cutaneous sclerosis

The main purpose is to evaluate the efficacy of SVF injections in the fingers of patients suffering from SSc on the Cochin hand functional scale evaluated at 12 months, in comparison to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Systemic Sclerosis ( limited or diffuse cutaneous shape)
* Men and women of more than 18 years old
* Patients wishing for a therapeutic alternative
* Functional Disability of the dominant hand authenticated by a functional index of the hand of Cochin functional scale upper to 20

Exclusion Criteria:

* Body mass index (weight in kilograms divided by height in meters squared) lower than 18
* Finger infection (including infected ulcer, ulcer with signs of local inflammation and clinical suspicion of osteitis)
* Contraindication to surgery
* Prescription of a new systemic treatment for SSc in the month before the inclusion Subjects infected with HIV, HCV ( hepatitis C virus) , HBV (hepatitis B virus), HTLV ( human T-cell leukemia virus) and syphilis
* Pre-menopausal women of reproductive age, taking no contraceptive method
* Patients receiving immunosuppressive therapy not including corticosteroid therapy < 10 mg/D and methotrexate

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2017-01; Primary Completion 2019-01 (Estimated); Study Completion 2019-08 (Estimated)

PRIMARY OUTCOMES:
Cochin hand functional scale | 12 months

SECONDARY OUTCOMES:
the severity (frequency and intensity of crises) of Raynaud's phenomenon | 12 months
the strength (Jamar et Pinch test) | 12 months
the trouble trophicity (health assesment questionnaire) | 12months
the pain in the hands (EVA pain scale), | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: catherine GEINDRE, Study Director — ASSISTANCE PUBLIQUE HOPITAUX MARSEILLE; BRIGITTE GRANEL, Principal Investigator — ASSISTANCE PUBLIQUE HOPITAUX MARSEILLE
Locations (1):
- Assistance Publique Hopitaux de Marseille, Marseille, France